CLINICAL TRIAL: NCT02777177
Title: Ecological Momentary Assessment of Behavioral and Psychosocial Predictors of Weight Loss Following Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, John Graham Thomas, Associate Professor (Research), The Miriam Hospital
Other Study IDs: R01DK108579 (NIH)
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Bariatric surgery is a powerful tool for producing significant and durable weight loss. Yet, not all patients achieve initial weight loss success and many patients have weight regain as early as 1-2 years post-surgery. Suboptimal weight loss patterns not fully explained by surgical, demographic, and medical factors has led to greater emphasis on patient behaviors evidenced by clinical guidelines that focus on appropriate eating and physical activity. However, research to inform such guidelines typically has relied on imprecise measures or not been specific to bariatric surgery. There is also little understanding of mechanisms by which psychosocial factors influence outcomes. Thus, there is a need to: (a) measure behaviors and psychosocial factors thought to be related to surgical outcomes (particularly those emphasized in guidelines) using innovative strategies to maximize data quality, (b) determine which behaviors and psychosocial factors are related to outcomes, and (c) explore how psychosocial factors influence weight both directly and via influences on behavior. Our research team was the first to employ innovative mobile health (mHealth) technology within an Ecological Momentary Assessment (EMA) framework to measure adherence to recommended behaviors at 6 months post-surgery. The investigators propose to build on this work by using EMA to measure behavioral, psychosocial, and environmental factors over a longer period to understand how they predict success and risk after surgery. An NIH-funded multi-sensor PiLR HEALTH platform will integrate objective sensor data measuring behaviors and the environments in which they are performed with self-report information collected via smartphone in real-time and in patients' natural environment. Participants (N=100) recruited from 2 ASMBS-designated centers of excellence will complete a 10-day EMA protocol pre-surgery and at 3, 6, and 12 months post-surgery to assess recommended behaviors [e.g., meal frequency, PA], psychosocial indicators with the most prior evidence of an association with surgical outcomes (e.g., mood/depression), and key environmental factors (e.g., type/quality of the food environment). Participants will also be weighed at the above time points. Along with describing patterns in behaviors and their relation to weight loss, the investigators will test causal models to understand how complex systems of behavioral, psychosocial, and environmental factors affect weight loss, and to identify optimal targets for intervention. This project has the potential to build a much more sophisticated and valid understanding of who is and is not successful after bariatric surgery and why. This new understanding will directly contribute to improved (i.e., specific, consistent, and validated) guidelines for recommended pre and postoperative behaviors, which could lead to improved surgical outcomes. The enhanced understanding will also inform behavioral, psychosocial, and environmental targets for intervention that are mostly likely to improve surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of at least 35 kg/m-squared

Exclusion Criteria:

* Currently involved in a weight loss or related behavioral form of treatment outside the context of standard surgical care
* Any condition that in the opinion of the investigators would preclude adherence to the measurement protocol, including plans to relocate, substance abuse or other significant psychiatric problems, or terminal illness

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with obesity who plan to have bariatric surgery within 8 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 12-months post bariatric surgery

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Miriam Hospital Weight Control and Diabetes Resarch Center, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bond DS, Smith KE, Schumacher LM, Vithiananthan S, Jones DB, Papasavas P, Webster J, Thomas JG. Associations of daily weight management-focused social support with weight loss, activity behaviors, and eating regulation in the context of metabolic and bariatric surgery. Obes Sci Pract. 2023 Nov 10;10(1):e717. doi: 10.1002/osp4.717. eCollection 2024 Feb. PMID 38263993
- [Derived] Goldstein SP, Thomas JG, Vithiananthan S, Blackburn GA, Jones DB, Webster J, Jones R, Evans EW, Dushay J, Moon J, Bond DS. Multi-sensor ecological momentary assessment of behavioral and psychosocial predictors of weight loss following bariatric surgery: study protocol for a multicenter prospective longitudinal evaluation. BMC Obes. 2018 Nov 5;5:27. doi: 10.1186/s40608-018-0204-6. eCollection 2018. PMID 30410772